CLINICAL TRIAL: NCT00345033
Title: Aripiprazole for Clozapine Associated Medical Morbidity
Brief Title: Effectiveness of Aripiprazole for Improving Side Effects of Clozapine in the Treatment of People With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David C. Henderson, Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01MH072635 (NIH); R01MH072635 (NIH); DSIR 83-ATAP
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Results first posted 2012-09-13 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia; Insulin Resistance
Keywords: Glucose Metabolism
MeSH Terms: conditions — Schizophrenia; Insulin Resistance | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will take aripiprazole 15mg/day for 8 weeks.
  Interventions: Drug: Aripiprazole
- 2 (Placebo Comparator): Participants will take placebo for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — 15-mg dose once a day for 8 weeks
  Arms: 1
Drug: Placebo — 1 tablet placebo dose once a day for 8 weeks
  Arms: 2

SUMMARY:
This study will evaluate the effects of combination treatment with aripiprazole and clozapine on insulin resistance, blood fat levels, and weight gain in people diagnosed with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a severely disabling brain disorder. People with schizophrenia often experience hallucinations and delusions, as well as overall difficulty with everyday functioning. Although the medications available to treat the disorder are generally effective, many cause undesirable side effects. Clozapine, for example, is a strong tranquilizer that functions like an antipsychotic medication. It has been shown to be effective in reducing the symptoms of schizophrenia, but can bring about serious side effects, including heart failure, weight gain, and diabetes. Aripiprazole, an atypical antipsychotic medication, has been shown to have fewer side effects than older antipsychotic drugs. The addition of aripiprazole to a clozapine treatment regimen may reduce the negative side effects of clozapine. This study will evaluate the effects of combination treatment with aripiprazole and clozapine on insulin resistance, blood fat levels, and weight gain in people with schizophrenia.

Individuals interested in participating in this 8-week, double-blind study will first attend a screening session at the study site. Medical and psychiatric evaluations will be completed, blood samples will be taken, and an EKG will be performed. Eligible participants will undergo baseline assessments and then be randomly assigned to receive either aripiprazole or placebo in addition to their prescribed dose of clozapine. Participants will take one 15-mg capsule of their assigned medication once a day for 8 weeks. Study visits will occur biweekly for the first 8 weeks, followed by one final follow-up visit at Week 12. At each study visit, medication will be distributed, and the following criteria will be assessed: vital signs; weight; complete blood count; medication side effects; and extrapyramidal symptoms (EPS), which are potential neurological side effects of antipsychotic medications and may include involuntary movements, tremors, and rigidity. The Week 8 visit will include an EKG, and assessments of the following criteria: vital signs; medication side effects; treatment efficacy; blood counts; weight and height; and waist and hip circumference. At baseline and Week 8, participants will also undergo a frequently sampled intravenous glucose tolerance test (FSIVGTT). This involves intravenous infusion of glucose followed by frequent blood sampling to measure insulin and glucose concentrations. During the 4 days prior to each FSIVGTT, participants will record their food intake and wear an activity monitor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia (any subtype) or schizoaffective disorder (any subtype)
* Treatment with clozapine for at least 1 year
* Stable dose of clozapine for at least 1 month
* Well established compliance with outpatient medications
* Female participants of non-childbearing potential or of childbearing potential and willing to practice appropriate birth control methods (complete abstinence from sexual intercourse, female sterilization, sterilization of male partner, implants of levonorgestrel, injectable progestogen, oral contraceptives, intrauterine devices, or double barrier methods of contraception using spermicide with either a condom or diaphragm) during the study

Exclusion Criteria:

* Current substance abuse
* Psychiatrically unstable
* Significant medical illness, including severe cardiovascular, hepatic, or renal disease
* History of immunosuppression
* Current or recent radiation or chemotherapy treatment for cancer
* Chronic use of steroids
* Pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-03; Primary Completion 2009-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C. Henderson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Schizophrenia Program, Boston, Massachusetts, United States

REFERENCES:
- [Background] Casey DE, Carson WH, Saha AR, Liebeskind A, Ali MW, Jody D, Ingenito GG; Aripiprazole Study Group. Switching patients to aripiprazole from other antipsychotic agents: a multicenter randomized study. Psychopharmacology (Berl). 2003 Apr;166(4):391-9. doi: 10.1007/s00213-002-1344-3. Epub 2003 Feb 28. PMID 12610718
- [Background] Goldstein LE, Sporn J, Brown S, Kim H, Finkelstein J, Gaffey GK, Sachs G, Stern TA. New-onset diabetes mellitus and diabetic ketoacidosis associated with olanzapine treatment. Psychosomatics. 1999 Sep-Oct;40(5):438-43. doi: 10.1016/S0033-3182(99)71210-7. No abstract available. PMID 10479950
- [Background] Hadigan C, Miller K, Corcoran C, Anderson E, Basgoz N, Grinspoon S. Fasting hyperinsulinemia and changes in regional body composition in human immunodeficiency virus-infected women. J Clin Endocrinol Metab. 1999 Jun;84(6):1932-7. doi: 10.1210/jcem.84.6.5738. PMID 10372689
- [Background] Henderson DC, Cagliero E, Gray C, Nasrallah RA, Hayden DL, Schoenfeld DA, Goff DC. Clozapine, diabetes mellitus, weight gain, and lipid abnormalities: A five-year naturalistic study. Am J Psychiatry. 2000 Jun;157(6):975-81. doi: 10.1176/appi.ajp.157.6.975. PMID 10831479
- [Background] Marder SR, McQuade RD, Stock E, Kaplita S, Marcus R, Safferman AZ, Saha A, Ali M, Iwamoto T. Aripiprazole in the treatment of schizophrenia: safety and tolerability in short-term, placebo-controlled trials. Schizophr Res. 2003 Jun 1;61(2-3):123-36. doi: 10.1016/s0920-9964(03)00050-1. PMID 12729864
- [Background] Visser M, Fuerst T, Lang T, Salamone L, Harris TB. Validity of fan-beam dual-energy X-ray absorptiometry for measuring fat-free mass and leg muscle mass. Health, Aging, and Body Composition Study--Dual-Energy X-ray Absorptiometry and Body Composition Working Group. J Appl Physiol (1985). 1999 Oct;87(4):1513-20. doi: 10.1152/jappl.1999.87.4.1513. PMID 10517786
- [Background] Wirshing DA, Boyd JA, Meng LR, Ballon JS, Marder SR, Wirshing WC. The effects of novel antipsychotics on glucose and lipid levels. J Clin Psychiatry. 2002 Oct;63(10):856-65. doi: 10.4088/jcp.v63n1002. PMID 12416594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Freedom Trail Clinic at the Erich Lindemann Mental Health Center and were studied at the General Clinical Research Center (GCRC) at the Massachusetts General Hospital (MGH), Boston and the Freedom Trail Clinic.
Pre-assignment Details: After providing written informed consent, subjects underwent a diagnostic evaluation by a research psychiatrist using the Structured Clinical Interview for DSM-IV (SCID). All subjects were screened and enrolled based on eligibility criteria. Baseline study assessments were completed prior to intervention.
Groups:
- Aripiprazole: Participants will take aripiprazole for 8 weeks.
- Placebo: Participants will take placebo for 8 weeks.
Period: Overall Study
Arm/Group | Aripiprazole | Placebo
Started | 20 | 18
Completed | 16 | 14
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Placebo | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 18 | 38
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (8.2) | 44.2 (8.9) | 44.25 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 16 | 10 | 26
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Cholesterol
Description: A comparison of aripiprazole group and placebo group in change in total cholesterol measured at Baseline and Week 8.
Time Frame: Measured at Baseline and Week 8
Population: The number of participants for analysis (intent to treat) were those that completed the study (N = 30).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 16 | 14
mg/dL | -15.3 (33.3) | 5.6 (34.0)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Non-Inferiority or Equivalence — A priori power calculation determined the power to detect a change in total cholesterol is over 99%; p = 0.125, ANCOVA

2. Primary Outcome: Change in Weight
Description: A comparison between aripiprazole group and placebo group in change in weight measured at Baseline and Week 8.
Time Frame: Measured at Baseline and Week 8
Population: The number of participants for analysis (intent to treat) were those that completed the study (N=30).
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 16 | 14
kg | -1.5 (2.3) | 0.3 (2.3)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Non-Inferiority or Equivalence — A priori power calculation determined the power to detect a change in weight will be over 99%; p = 0.109, ANCOVA

3. Primary Outcome: Change in Body Mass Index (BMI)
Description: A comparison between aripiprazole group and placebo group of change in Body Mass Index (BMI) measured at Baseline and Week 8.
Time Frame: Measured at Baseline and Week 8
Population: The number of participants for analysis (intent to treat) were those that completed the study (N=30).
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 16 | 14
kg/m^2 | -0.52 (0.79) | 0.03 (0.85)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Non-Inferiority or Equivalence — A priori power calculation determined the power to detect a change in Body Mass Index (BMI) will be over 99%; p = 0.229, ANCOVA

4. Primary Outcome: Change in Glucose Metabolism
Description: A comparison between the aripiprazole group and placebo group in change in glucose metabolism measured at Baseline and Week 8.
Time Frame: Measured at Baseline and Week 8
Population: The number of participants for analysis (intent to treat) were those that completed the study (N=30).
Measure: Mean (Standard Deviation); unit: min^-1
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 16 | 14
min^-1 | 0.003 (0.006) | -0.005 (0.007)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Non-Inferiority or Equivalence — A priori power calculation determined the power to detect a change in glucose metabolism to be 90%; p = 0.010, ANCOVA

5. Primary Outcome: Change in Triglycerides
Time Frame: Measured at Baseline and Week 8
Population: The number of participants for analysis (intent to treat) were those that completed the study (N=30)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 16 | 14
mg/dL | -5.9 (75.1) | -7.3 (100.3)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Non-Inferiority or Equivalence — A priori power calculation determined the power to detect a change in triglycerides will be 81%; p = 0.982, ANCOVA

6. Primary Outcome: Change in Insulin Resistance
Description: A comparison between aripiprazole group and placebo group of change in insulin resistance measured at Baseline and Week 8.
Time Frame: Measured at Baseline and Week 8
Population: The number of participants for analysis (intent to treat) were those that completed the study (N=30)
Measure: Mean (Standard Deviation); unit: HOMA score
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 16 | 14
HOMA score | 0.6 (3.8) | 0.65 (1.9)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Non-Inferiority or Equivalence — A priori power calculation determined the power to detect a change in Insulin Resistance will be 90%; p = 0.082, ANCOVA

ADVERSE EVENTS:
Arm/Group | Aripiprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 4/16 | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=16) | Placebo (N=14)
dizziness during IVGTT procedure (General disorders) | 0 (0) | 1 (1) — Subject experienced dizziness and hunger during IVGTT procedure. He was given orange juice and food, and the symptoms had resolved by the time he left the hospital. Coordinator contacted subject later that afternoon who reported feeling fine.
eye irritation/swelling (Eye disorders) | 1 (1) | 0 (0) — Subject visited Mass Eye and Ear with eye swelling and irritation. He was given Visine Tears after which the swelling and irritation resolved.
psychiatric decompensation (Psychiatric disorders) | 1 (1) | 0 (0) — Subject stayed at McLean Hospital for psychiatric evaluation over 1 night. His medications were not changed. He was seen by his psychiatrist 6 days later who confirmed that subject was doing well. Subject was admitted prior to any study procedures.
asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Subject experienced asthma attack. Subject has a history of asthma. Subject was given two nebulizer treatments at urgent care, which resolved the symptom, and she was released the same night. Subject was proscribed Adviar.
stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Subject called ambulance for stomach pain. She was given Maalox at the ER, which resolved the symptom, and she was discharged.
psychiatric decompensation (Psychiatric disorders) | 1 (1) | 0 (0) — Subject was hospitalized at BI after worsening psychiatric symptoms. It was discovered that subject was taking a lesser dosage than proscribed of his antipsychotic. Subject's dosage was adjusted and he was released.
psychiatric decompensation (Psychiatric disorders) | 1 (1) | 0 (0) — Subject stopped taking all of his medications including study medication, and was hospitalized after worsening psychiatric symptoms. Subject was terminated from the study.

LIMITATIONS AND CAVEATS:
The limitations of this study include the relatively small sample size, short intervention period (8 weeks) and the lack of generalizability of our findings to patients with schizophrenia treated by antipsychotic agents other than clozapine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes